CLINICAL TRIAL: NCT05912725
Title: Evaluation of the Accuracy of Conventional and Digital Implant Impression Techniques in Bilateral Distal Extension Cases
Brief Title: Conventional Impressions Versus Digital Impression Techniques for Implant Supported Screw Retained Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Wafaa elashry, Assistant lecturer at prosthodontic department, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-9-20-1
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Partial Edentulism Class 1
Keywords: Digital impression; implant impression; impression accuracy; Digital work flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accuracy of Implant impression techniques (Experimental): Active comparative : digital implant impression Participants underwent intra-oral scanning digital impression
  Experimental : conventional implant impression Participants underwent conventional impressions And right side of pt mouth received screw retained prosthesis constructed from conventional impression left side received screws retained prosthesis constructed from digital impression
  Interventions: Procedure: Implant placement

INTERVENTIONS:
Procedure: Implant placement — 4 implants were placed , 2 implants in each side of the patient mouth opposite lower second premolar and second molar
  4 implants were placed , 2 implants in each side of the patient mouth opposite lower second premolar and second molar

SUMMARY:
The purpose was to evaluate the accuracy of traditional and digital implant level impression procedures by using three-dimensional superimposition analysis , and evaluate the passive fit of screw- retained implant supported restorations fabricated using conventional and digital impression techniques in bilateral distal extension cases (class I kennedy classification)

DETAILED DESCRIPTION:
Eight patients who had missing all mandibular posterior teeth except first premolars were included in this study. In each patient, 4 implants were placed, 2 in each side to support 3 units screw retained zirconia restorations. Three months after implant placement, each patient underwent two implant level impression techniques (n=8) for each technique: Conventional implant impressions CII (pick-up, splinted transfers), and digital implant impressions DII were captured with TRIOS 3 Shape intraoral optical scanner. In this study, digital impression was considered as a reference data.

ELIGIBILITY:
Inclusion Criteria:

* All participants have sufficient bone length and width for implant insertion.
* General health of the patients was evaluated by taking a full medical history to ensure that these patients were free from any systemic conditions that would have impaired implant osseointegration
* Good oral hygiene
* Sufficient inter-arch spaces
* The opposing arch was almost dentulous, and any missing teeth were restored using a fixed partial denture.

Exclusion Criteria:

* parafunctional habits
* Heavy smoking
* Those patients with systemic diseases that may influence soft or hard tissue healing.
* Patients with a history of radiation therapy in the head and neck region.
* Patients with a history of radiation therapy in the head and neck region.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of digital and conventional implant impression techniques in partially edentulous patient | 12 months
  GOM Inspect 2016, Gom GmbH,) that was used to superimpose the Standard tessellation language (STL) datasets of conventional open tray impression technique onto the STL file of the reference (digital implant impression technique) to assess the accuracy and calculate the three-dimensional deviations of scan bodies in color- coding map in micrometers (µm)

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa Y El ashry, MSc, Principal Investigator — Tanta university ,Faculty of Dentistry, Prosthodontics department; Wafaa Y El ashry, Principal Investigator — Tanta university, Faculty of Dentistry, Prosthodontics department; Wafaa Y El ashry, MSc, Principal Investigator — Tanta University
Locations (1):
- Wafaa youssif El ashry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elashry WY, Elsheikh MM, Elsheikh AM. Evaluation of the accuracy of conventional and digital implant impression techniques in bilateral distal extension cases: a randomized clinical trial. BMC Oral Health. 2024 Jul 5;24(1):764. doi: 10.1186/s12903-024-04495-0. PMID 38970004